CLINICAL TRIAL: NCT03554460
Title: Evaluation of Carbon-dioxide Rebreathing During Exercise With the Increasing Ventilation Assisted by Noninvasive Ventilation With a Dual-limb Circuit
Brief Title: Evaluation of CO2 Rebreathing During Exercise With the Increasing Ventilation Assisted by NIV With a Dual-limb Circuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yonger Ou, Principal Investigator, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIRD201802
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dual-limb NIV (Experimental): A maximal cycle exercise test with the participants assisted by BiPAP (Servo i, Maquet, Siemens) receiving 10 cmH2O pressure support in addition to oxygen therapy. During the test, breathing pattern, inspiratory flow of the inhalation limb and expiratory flow of the exhalation limb, fractional concentration of inspired CO2 (FiCO2) of the inspiratory line was measured for each breath were recorded.
  Interventions: Device: dual-limb NIV

INTERVENTIONS:
Device: dual-limb NIV — dual-limb NIV was served with servo i ventilator

SUMMARY:
Ventilated by a single-limb tubing with PEV caused CO2 rebreathing to COPD patients during exercise with the increasing ventilation. The aim of this study was to evaluate whether CO2 rebreathing could be avoided with the use of the dual-limb circuit, to provide a theoretical basis of more rational clinical application of NIV in the setting of increasing ventilation(eg, after exercise).

DETAILED DESCRIPTION:
Exercise training is a key component of pulmonary rehabilitation. It has shown signifcant improvements in both exercise tolerance and quality of life in patients with COPD. The intensity of exercise training is of great importance to yield a true physiologic effect. However, in patients with severe COPD, exertional dyspnea and leg fatigue make it impossible for the patient to maintain intensity of training for enough time to achieve a physiologic training effect. NIV has been reported to be used as support for exercise to improve exercise tolerance and respiratory performances in patients with mild-to-severe COPD with inconsistent results. Evidence from previous studies have suggested that NIV with a single-limb circuit with Whisper Swivel II expiratory valve or Plateau exhalation valve assisted during exercise in patients with COPD caused CO2 rebreathing. CO2 rebreathing may have a negative impact on efficacy. Previous studies have proved that exercise tolerance was improved ventilated by NIV with a dual-limb circuit. In theory, NIV with a dual-limb circuit consists of one inhalation limb that introduces air into the patient's airways and one exhalation limb that leads exhaled gas outside of the airways, there is no risk of rebreathing. However, there was no report on whether there's no risk of rebreathing in COPD patients ventilated during exercise by a dual-limb circuit. Therefore, the aim of the study was to determine whether there was no CO2 rebreathing occurred assisted with NIV with dual-limb circuit in patients with stable severe COPD after exercise with exertional dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* presented clinically stable (no exacerbation in the 4 weeks prior to study
* participation or with no change in medications);
* physician diagnosed COPD, forced expiratory volume in 1s (FEV1) < 50% predicted; dyspnea as a main symptom that limited daily activities.

Exclusion Criteria:

* subjects with obvious pulmonary bullae demonstrated by chest CT scan or X-ray; examination or facial trauma/malformation, recent facial, upper airway or upper gastrointestinal tract surgery, that would preclude receiving NIV therapy;
* a history of coronary artery disease or cardiac arrhythmias or potential electrocardiographic alterations;
* a history of uncontrolled hypertension, or other respiratory diseases;
* patients with musculoskeletal or neurological disorders;
* failure to comply with the research protocol.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
fractional concentration of inspired CO2 | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
  FiCO2

SECONDARY OUTCOMES:
inspiratory flow of the inhalation limb | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
  Vti/Ti
expiratory flow of the exhalation limb | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
  Vte/Te
breathing pattern | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
  Ti、Te、Ti/Ttot、RR

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, Study Director — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China